CLINICAL TRIAL: NCT00006184
Title: Active Immunization of Sibling Stem Cell Transplant Donors Against Purified Myeloma Protein of the Stem Cell Recipient With Multiple Myeloma in the Setting of Non-Myeloablative, HLA-Matched Allogeneic Peripheral Blood Stem Cell Transplantation
Brief Title: Chemotherapy, Stem Cell Transplantation and Donor and Patient Vaccination for Treatment of Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ronald Gress, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 000201; 00-C-0201; NCT00020306 (obsolete NCT alias)
Record Dates: First submitted 2000-08-23; First posted 2000-08-24 (Estimated); Results first posted 2013-01-24 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-09

CONDITIONS: Multiple Myeloma
Keywords: Immunoablative; Mobilization; Apheresis; Multiple Myeloma; IgG Multiple Myeloma; IgA Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Cyclophosphamide; Cyclosporine; Doxorubicin; Etoposide; fludarabine phosphate; Prednisone; Vincristine; Methotrexate; Colony-Stimulating Factors; Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Recipient - Chemotherapy Group (Experimental): Induction chemotherapy with fludarabine, etoposide, doxorubicin, vincristine, cyclophosphamide, prednisone, and granulocyte colony stimulating factor (GCSF) followed by transplant preparative regimen chemotherapy with fludarabine, cyclophosphamide, mesna, cyclosporine, and methotrexate, followed by stem cell infusion and immunization.
  Interventions: Drug: Bortezomib; Drug: Cyclophosphamide; Drug: Cyclosporine; Drug: Doxorubicin hydrochloride; Drug: Etoposide; Drug: Fludarabine phosphate; Drug: Prednisone; Drug: Vincristine Sulfate; Drug: Methotrexate; Biological: GCSF (granulocyte colony stimulating factor)
- Donor - Vaccine Generation Group (Other): 3 subcutaneous injections of myeloma protein within 10 weeks before stem cell collection. The first (week 0) second (week 2), and third injection (week 6) with Id-KLH (Anti-idiotype-keyhole limpet hemocyanin) (0.5 mg subcutaneous day 1) and Granulocyte macrophage-colony stimulating factor (GM-CSF) (250 mcg/m^2 subcutaneous on days 1-4). Stem cell collection is 4 weeks after the third vaccination.
  Interventions: Drug: Myeloma Immunoglobulin Idiotype Vaccine; Drug: Bortezomib; Biological: GMCSF (granulocyte macrophage colony stimulating factor)

INTERVENTIONS:
Drug: Myeloma Immunoglobulin Idiotype Vaccine — 3 subcutaneous (SC) injections of myeloma protein within 10 weeks before stem cell collection the first (week 0), second (week 2), and third injection (week 6) with Id-KLH (0.5 mg SC day 1)
  Arms: Donor - Vaccine Generation Group
Drug: Bortezomib — Induction chemotherapy: 1.3 mg/m^2 bolus intravenous injection twice weekly for 2 weeks (days 1, 4, 8, 11) followed by 10 day rest period (day 12-21)
  Other Names: Velcade; PS341
Drug: Cyclophosphamide — Induction chemotherapy: 600 mg/m^2 day 4 Transplant: 1200 mg/m^2 intravenous x 4 days (days -6, -5, -4, -3)
  Other Names: Cytoxan; CTX
  Arms: Recipient - Chemotherapy Group
Drug: Cyclosporine — Transplant: 2 mg/kg intravenous every 12 hours continuous intravenous or by mouth (PO) until day + 180
  Other Names: Sandimmune; Cyclosporin A
  Arms: Recipient - Chemotherapy Group
Drug: Doxorubicin hydrochloride — Induction chemotherapy: 10 mg/m^2 day continuous intravenous (CIV) days 1-3
  Arms: Recipient - Chemotherapy Group
Drug: Etoposide — Induction chemotherapy: 50 mg/m^2 day continuous intravenous days 1-3
  Other Names: Vepesid
  Arms: Recipient - Chemotherapy Group
Drug: Fludarabine phosphate — Induction chemotherapy: 25 mg/m^2 day intravenous days 1-3 Transplant: 30 mg/m^2 day x 4 days (days -6, -5, -4, -3 )
  Other Names: Fludara
  Arms: Recipient - Chemotherapy Group
Drug: Prednisone — 60 mg/m^2 day 1-4
  Other Names: Deltasone
  Arms: Recipient - Chemotherapy Group
Drug: Vincristine Sulfate — Induction chemotherapy: 0.5 mg/m^2 day continuous intravenous days 1-3
  Arms: Recipient - Chemotherapy Group
Drug: Methotrexate — Transplant: 5 mg/m^2 intravenous on days +1, +3, +6, +11
  Other Names: MTX; Methotrexate sodium
  Arms: Recipient - Chemotherapy Group
Biological: GMCSF (granulocyte macrophage colony stimulating factor) — 250 mcg/m^2 subcutaneously every day, days 1-4
  Arms: Donor - Vaccine Generation Group
Biological: GCSF (granulocyte colony stimulating factor) — 10 mcg/kg per day subcutaneously daily from day 5 until absolute neutrophil count (ANC) > 1000/ul x 2 days
  Other Names: Filgrastim; Neupogen
  Arms: Recipient - Chemotherapy Group

SUMMARY:
Background:

The mainstay of therapy for newly diagnosed multiple myeloma patients remains systemic chemotherapy. Although partial remissions of up to 60% are obtained with conventional regimens, multiple myeloma is essentially an incurable disease with a median survival of approximately 30 months.

Allogeneic stem cell transplantation (SCT) results in a high percentage of complete remissions, but it can be associated with significant treatment-related mortality, which has been primarily attributed to conventional myeloablative transplant regimens.

Recent clinical studies have shown that highly immunosuppressive yet non-myeloablative doses of fludarabine-based chemotherapy can result in alloengraftment. Even with a reduction in treatment related mortality, success with allogeneic SCT is limited by a significant risk of relapse.

Donor immunization with myeloma Id in the setting of a non-myeloablative allogeneic SCT may represent a novel strategy for the treatment of multiple myeloma.

Objectives:

Primary Objectives:

To induce cellular and humoral immunity in allogeneic stem cell donors and recipients against the unique idiotype expressed by the recipient's myeloma.

To determine whether antigen-specific immunity, induced in the stem cell donor, can be passively transferred to the allogeneic SCT recipient in the setting of a non-myeloablative conditioning regimen.

Secondary Objectives:

To evaluate the effect of the Fludarabine-(etoposide, doxorubicin, vincristine, prednisone, cyclophosphamide) EPOCH regimen on host T cell depletion and myeloid depletion prior to allogeneic SCT.

To determine the efficacy of a novel conventional chemotherapy regimen (Fludarabine-EPOCH) in the setting multiple myeloma.

To determine the treatment-related morbidity and mortality of allogeneic stem cell transplantation using a non-myeloablative conditioning regimen in multiple myeloma.

To determine if the re-vaccination of allogeneic stem cell donors with the unique idiotype expressed by the recipient's myeloma will enhance cellular and humoral immunity to patient specific-idiotype prior to lymphocyte donation for the treatment of patients with recurrent or progressive disease after transplantation.

Eligibility:

Patients 18-75 years of age with Immunoglobulin G (IgG) or Immunoglobulin A (IgA) multiple myeloma.

Patients must have achieved at least a partial remission following initial conventional chemotherapy regimen or after autologous stem cell transplantation.

Consenting first degree relative matched at 6/6 or 5/6 human leukocyte antigen (HLA) antigens.

Design:

Phase 2 trial using a non-myeloablative conditioning regimen to reduce treatment-related toxicity.

Recipient will undergo a plasmapheresis to obtain starting material for the isolation of idiotype

protein. Donors would be immunized with an Id vaccine prepared from the patient.

Prior to transplantation patients would receive a conventional chemotherapy regimen which contains agents active in myeloma and is T cell depleting. The allogeneic SCT would be performed with a conditioning regimen consisting of cyclophosphamide and fludarabine. The stem cell source would be blood mobilized with filgrastim. Recipients will be immunized with the Id vaccine following transplantation.

DETAILED DESCRIPTION:
Background:

The mainstay of therapy for newly diagnosed multiple myeloma patients remains systemic chemotherapy. Although partial remissions of up to 60% are obtained with conventional regimens, multiple myeloma is essentially an incurable disease with a median survival of approximately 30 months.

Allogeneic stem cell transplantation (SCT) results in a high percentage of complete remissions, but it can be associated with significant treatment-related mortality, which has been primarily attributed to conventional myeloablative transplant regimens.

Recent clinical studies have shown that highly immunosuppressive yet non-myeloablative doses of fludarabine-based chemotherapy can result in allo-engraftment. Even with a reduction in treatment related mortality, success with allogeneic SCT is limited by a significant risk of relapse.

Donor immunization with myeloma Id in the setting of a non-myeloablative allogeneic SCT may represent a novel strategy for the treatment of multiple myeloma.

Objectives:

Primary Objectives:

To induce cellular and humoral immunity in allogeneic stem cell donors and recipients against the unique idiotype expressed by the recipient's myeloma.

To determine whether antigen-specific immunity, induced in the stem cell donor, can be passively transferred to the allogeneic SCT recipient in the setting of a non-myeloablative conditioning regimen.

Secondary Objectives:

To evaluate the effect of the Fludarabine-EPOCH regimen on host T cell depletion and myeloid depletion prior to allogeneic SCT.

To determine the efficacy of a novel conventional chemotherapy regimen (Fludarabine-EPOCH) in the setting multiple myeloma.

To determine the treatment-related morbidity and mortality of allogeneic stem cell transplantation using a non-myeloablative conditioning regimen in multiple myeloma.

To determine if the re-vaccination of allogeneic stem cell donors with the unique idiotype expressed by the recipient's myeloma will enhance cellular and humoral immunity to patient specific-idiotype prior to lymphocyte donation for the treatment of patients with recurrent or progressive disease after transplantation.

Eligibility:

Patients 18-75 years of age with IgG or IgA multiple myeloma.

Patients must have achieved at least a partial remission following initial conventional chemotherapy regimen or after autologous stem cell transplantation.

Consenting first degree relative matched at 6/6 or 5/6 HLA antigens.

Design:

Phase 2 trial using a non-myeloablative conditioning regimen to reduce treatment-related toxicity.

Recipient will undergo a plasmapheresis to obtain starting material for the isolation of idiotype protein. Donors would be immunized with an Id vaccine prepared from the patient.

Prior to transplantation patients would receive a conventional chemotherapy regimen which contains agents active in myeloma and is T cell depleting. The allogeneic SCT would be performed with a conditioning regimen consisting of cyclophosphamide and fludarabine. The stem cell source would be blood mobilized with filgrastim. Recipients will be immunized with the Id vaccine following transplantation.

ELIGIBILITY:
* INCLUSION CRITERIA: Collection of plasma in recipient:

Patients with Immunoglobulin G (IgG) or Immunoglobulin A (IgA) multiple myeloma.

Patients have siblings.

Human leukocyte antigen (HLA) typing of recipient and donor(s) initiated.

Viral antibody screening initiated.

INCLUSION CRITERIA: Recipient:

Patients with IgG or IgA multiple myeloma.

Patients must have achieved at least a partial remission following initial conventional chemotherapy regimen or after autologous stem cell transplantation. Patients who have undergone tandem autologous stem transplants are eligible if they meet all other eligibility criteria. Patients who have achieved at least a partial remission to initial (primary) conventional chemotherapy will be encouraged to proceed to autologous transplantation, but will also be eligible for this protocol.

Patients 18-75 years of age. The upper age limit was chosen as it is felt that the toxicities would exceed potential benefit in this older population.

Karnofsky performance status greater than or equal to 80%.

Life expectancy greater than 6 months.

Left ventricular ejection fraction has to be greater than 50% by either multi-gated acquisition scan (MUGA) or 2-D echo.

Carbon monoxide diffusing capacity (DLCO) greater than 50% of the expected value when corrected for hemoglobin (Hb)(96).

Creatinine less than or equal to 1.5 mg/dl and a creatinine clearance greater than or equal to 50 ml/min.

Direct bilirubin less than or equal to 2.0 mg/dl serum glutamic oxaloacetic transaminase (SGOT) less than 4x top normal.

M-protein: the concentration in the harvested plasma must be greater than 70% of the total Ig of the corresponding isotype.

Patients must be human immunodeficiency virus (HIV)-negative. There is the theoretical possibility that the degree of immune suppression associated with the treatment may result in progression of HIV infection. Patients may be Hepatitis B core antigen positive, but surface antigen negative and without evidence of active infection. Patients must be Hepatitis C negative.

Not pregnant or lactating. Patients of childbearing potential must use an effective method of contraception. The effects of the chemotherapy, the subsequent transplant and the medications used after the transplant are highly likely to be harmful to a fetus. The effects upon breast milk are also unknown and may potentially be harmful to the infant.

Consenting first degree relative matched at 6/6 or 5/6 HLA antigens, this may include a mismatch at the D locus.

Ability to give informed consent.

INCLUSION CRITERIA: Donor:

Age 18-75 years. As the potential cerebrovascular and cardiac complications may potentially increase with age, age 75 has been chosen arbitrarily as the upper age limit. However, if it is determined after initial accrual of patients in this upper age range that this procedure is relatively safe, the age range may be extended.

No physical contraindications to stem cell donation (i.e. severe atherosclerosis, auto-immune disease, cerebrovascular accident, active malignancy (97). Patients with severe atherosclerosis by history will receive a cardiology consult and be judged eligible on a case by case basis.

Donors must be HIV-negative, hepatitis B surface antigen (HBsAg-), and Hepatitis C antibody negative. This is to prevent the possible transmission of these infections to the recipient.

Not pregnant or lactating. Donors of childbearing potential must use an effective method of contraception. The effects of cytokine administration on a fetus are unknown and may be potentially harmful. The effects upon breast milk are also unknown and may potentially be harmful to the infant.

Normal cluster of differentiation 4 (CD4) and cluster of differentiation 8 (CD8) numbers as defined by Clinical Center standards.

Ability to give informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2001-02-08 (Actual); Primary Completion 2008-01-12 (Actual); Study Completion 2008-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claude Sportes, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stevenson GT, Stevenson FK. Antibody to a molecularly-defined antigen confined to a tumour cell surface. Nature. 1975 Apr 24;254(5502):714-6. doi: 10.1038/254714a0. No abstract available. PMID 47617
- [Background] Stevenson GT, Elliott EV, Stevenson FK. Idiotypic determinants on the surface immunoglobulin of neoplastic lymphocytes: a therapeutic target. Fed Proc. 1977 Aug;36(9):2268-71. No abstract available. PMID 69552
- [Background] Miller RA, Maloney DG, Warnke R, Levy R. Treatment of B-cell lymphoma with monoclonal anti-idiotype antibody. N Engl J Med. 1982 Mar 4;306(9):517-22. doi: 10.1056/NEJM198203043060906. No abstract available. PMID 6173751
- [Result] Foglietta M, Neelapu SS, Kwak LW, Jiang Y, Nattamai D, Lee ST, Fowler DH, Sportes C, Gress RE, Steinberg SM, Vence LM, Radvanyi L, Dwyer KC, Qazilbash MH, Bryant RN, Bishop MR. Neoantigen and tumor antigen-specific immunity transferred from immunized donors is detectable early after allogeneic transplantation in myeloma patients. Bone Marrow Transplant. 2013 Feb;48(2):269-77. doi: 10.1038/bmt.2012.132. Epub 2012 Jul 9. PMID 22773122
- [Derived] Jamshed S, Fowler DH, Neelapu SS, Dean RM, Steinberg SM, Odom J, Bryant K, Hakim F, Bishop MR. EPOCH-F: a novel salvage regimen for multiple myeloma before reduced-intensity allogeneic hematopoietic SCT. Bone Marrow Transplant. 2011 May;46(5):676-81. doi: 10.1038/bmt.2010.173. Epub 2010 Jul 26. PMID 20661232

RESULTS

PARTICIPANT FLOW:
Groups:
- Recipient - Chemotherapy Group: Induction chemotherapy with fludarabine, etoposide, doxorubicin, vincristine, cyclophosphamide, prednisone, and granulocyte colony stimulating factor ( GCSF) followed by transplant preparative regimen chemotherapy with fludarabine, cyclophosphamide, mesna, cyclosporine, and methotrexate, followed by stem cell infusion and immunization.
- Donor - Vaccination Generation Group: 3 subcutaneous injections of myeloma protein within 10 weeks before stem cell collection. The first (week 0) second (week 2), and third injection (week 6) with Id-KLH (Anti-idiotype-keyhole limpet hemocyanin) (0.5 mg subcutaneous day 1) and Granulocyte macrophage-colony stimulating factor (GM-CSF) (250 mcg/m^2 subcutaneous on days 1-4). Stem cell collection is 4 weeks after the third vaccination
Period: Overall Study
Arm/Group | Recipient - Chemotherapy Group | Donor - Vaccination Generation Group
Started | 10 | 10
Completed | 9 | 10
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Recipient - Chemotherapy Group: Induction chemotherapy with fludarabine, etoposide, doxorubicin, vincristine, cyclophosphamide, prednisone, and GCSF followed by transplant preparative regimen chemotherapy with fludarabine, cyclophosphamide, mesna, cyclosporine, and methotrexate, followed by stem cell infusion and immunization.
- Donor - Vaccination Generation Group: 3 subcutaneous injections of myeloma protein within 10 weeks before stem cell collection. The first (week 0) second (week 2), and third injection (week 6) with Id-KLH (0.5 mg subcutaneous day 1) and Granulocyte macrophage-colony stimulating factor (GM-CSF) (250 mcg/m^2 subcutaneous on days 1-4). Stem cell collection is 4 weeks after the third vaccination
- Total: Total of all reporting groups
Arm/Group | Recipient - Chemotherapy Group | Donor - Vaccination Generation Group | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (4.59) | 50.8 (6.05) | 52. (5.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 7 | 4 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 8 | 16
  Hispanic | 1 | 1 | 2
  Non Hispanic | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Immune Response
Description: Immune cell depletion is defined as immunosuppression of participants T cells prior to transplant measured by cluster of differentiation 4 (CD4) counts (i.e. cells) > 50 cells per ul.Immune T-cell depletion helps to reduce the ability to reject allogeneic cells in participants and is required for engraftment. Engraftment is the body's ability to accept donor cells.
Time Frame: 105 days
Population: This outcome measure was only pre-specified to be measured in the recipient Arm/Group.
Measure: Number; unit: Particpants
Arm/Group | Recipient - Chemotherapy Group
Number analyzed (Participants) | 10
Particpants | 7

2. Primary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events see the adverse event module.
Time Frame: 9 years
Measure: Count of Participants; unit: Participants
Arm/Group | Recipient - Chemotherapy Group | Donor - Vaccination Generation Group
Number analyzed (Participants) | 10 | 10
Participants | 10 | 10

ADVERSE EVENTS:
Time Frame: 9 years
Arm/Group | Recipient - Chemotherapy Group | Donor - Vaccination Generation Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 10/10 | 0/10
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recipient - Chemotherapy Group (N=10) | Donor - Vaccination Generation Group (N=10)
Abdominal pain or cramping (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Diarrhea (without colostomy) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — (fever of unknown origin without clinically or microbiologically documented infection)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Infection without neutropenia (Infections and infestations) | 2 (2) | 0 (0)
Leukocytes (total WBC) (Investigations) | 6 (13) | 0 (0)
Leukocytes (total WBC) for BMT (Investigations) | 4 (4) | 0 (0)
Metabolic-Other (GGT) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Mood alteration::Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Nausea and vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neurologic-Other (Neuropathy) (Nervous system disorders) | 1 (1) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 7 (16) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) for BMT (Investigations) | 8 (10) | 0 (0)
Platelets (Investigations) | 2 (2) | 0 (0)
Platelets for BMT (Investigations) | 2 (2) | 0 (0)
SGOT (AST) (Investigations) | 1 (1) | 0 (0)
SGPT (ALT) (Investigations) | 2 (2) | 0 (0)
Transfusion: Platelets (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recipient - Chemotherapy Group (N=10) | Donor - Vaccination Generation Group (N=10)
Abdominal pain or cramping (Gastrointestinal disorders) | 2 (3) | 3 (3)
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Alkaline phosphatase (Investigations) | 3 (6) | 2 (2)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1) | 0 (0)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 2 (4) | 1 (1)
Allergy - Other (Transfusion reaction (platelets) (Immune system disorders) | 1 (1) | 0 (0)
Amylase (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Bilirubin (Investigations) | 4 (11) | 0 (0)
Bilirubin - graft versus host disease (GVHD) (Investigations) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 6 (17) | 3 (6)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Catheter-related infection (Infections and infestations) | 4 (5) | 0 (0)
Chest pain (non-cardiac and non-pleuritic) (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (5) | 1 (2)
Constitutional Symptoms-Other (CGVHD-skin) (General disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Creatinine (Investigations) | 7 (12) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (6) | 0 (0)
Diarrhea (with colostomy) (Gastrointestinal disorders) | 1 (2) | 0 (0)
Diarrhea (without colostomy) (Gastrointestinal disorders) | 7 (14) | 0 (0)
Diarrhea (without colostomy) BMT (Gastrointestinal disorders) | 1 (4) | 0 (0)
Dizziness/lightheadedness (Nervous system disorders) | 1 (1) | 2 (3)
Dyspareunia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
Edema (General disorders) | 2 (2) | 0 (0)
Erythema multiforme (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (3)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 6 (10) | 4 (5)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 8 (22) | 1 (3)
Flushing (Vascular disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (4)
Hemoglobin (hgb) (Investigations) | 10 (41) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemorrhage/bleeding without grade 3 or 4 thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (6) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (6) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 2 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 6 (6) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 6 (14) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (5) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (9) | 0 (0)
Ileus (or neuroconstipation) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutropenia (Infections and infestations) | 6 (9) | 0 (0)
Infection w/out neutropenia, catheter related (Infections and infestations) | 1 (1) | 0 (0)
Infection without neutropenia (Infections and infestations) | 6 (15) | 0 (0)
Infection without neutropenia, blood (Infections and infestations) | 1 (2) | 0 (0)
Infection without neutropenia, C-diff (Infections and infestations) | 1 (1) | 0 (0)
Infection without neutropenia, Nasal Pharynx (Infections and infestations) | 1 (1) | 0 (0)
Infection without neutropenia, wound (Infections and infestations) | 1 (3) | 0 (0)
Infection, Other (Upper respiratory infection (URI)) (Infections and infestations) | 1 (1) | 0 (0)
Infection: blood (Infections and infestations) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 8 (25) | 10 (29)
Injection site reaction, bilat arms (General disorders) | 1 (2) | 0 (0)
Injection site reaction, bilat legs (General disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Joint, muscle, or bone (osseous)- Other (Calf cramping) (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Leukocytes (total WBC) (Investigations) | 8 (34) | 0 (0)
Leukocytes (total WBC) for BMT (Investigations) | 4 (9) | 0 (0)
Lymphatics (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphatics-Other (Adenopathy) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphopenia (Investigations) | 7 (29) | 1 (1)
Metabolic-Other (Hyperbilirubinemia; hyperbilirubinemia r/t GVH) (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Mood alteration-depression (Psychiatric disorders) | 1 (1) | 0 (0)
Mood alteration-euphoria (Psychiatric disorders) | 1 (1) | 0 (0)
Myalgia (muscle ache) (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (7)
Nausea (Gastrointestinal disorders) | 9 (25) | 0 (0)
Neuropathic pain (Nervous system disorders) | 1 (1) | 0 (0) — (e.g., jaw pain, neurologic pain, phantom limb pain, post infection-infectious neuralgia, or painful neuropathies
Neuropathy-sensory (Nervous system disorders) | 5 (5) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 7 (19) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) for BMT (Investigations) | 4 (9) | 0 (0)
Ocular-Other (Ocular cGVHD) (Eye disorders) | 1 (1) | 0 (0)
Pain - Other (General disorders) | 4 (8) | 2 (3) — catheter site; hp and leg; hip and leg exacerbation related GCSF; meniscus tear
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Pigmentation changes (e.g., vitiligo) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Platelets (Investigations) | 7 (22) | 3 (4)
Platelets for BMT (Investigations) | 6 (11) | 0 (0)
Pleural effusion (non-malignant) (Psychiatric disorders) | 1 (1) | 0 (0)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pericardial effusion/pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 3 (3)
Pulmonary-Other (URI) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 6 (11) | 2 (2)
Rash/desquamation for BMT (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rectal bleeding/hematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rigors/chills (General disorders) | 2 (2) | 2 (4)
Salivary gland changes (Gastrointestinal disorders) | 1 (1) | 0 (0)
SGOT (AST) (Investigations) | 8 (42) | 2 (2)
SGPT (ALT) (Investigations) | 8 (32) | 3 (3)
Skin-Other (Drug reaction face, hands, neck) (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (General disorders) | 4 (5) | 0 (0)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) for BMT (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Taste disturbance (dysgeusia) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Thrombosis/embolism (Vascular disorders) | 1 (1) | 0 (0)
Transfusion: Platelets for BMT (Investigations) | 6 (6) | 0 (0)
Transfusion: pRBCs (Investigations) | 3 (4) | 0 (0)
Transfusion: pRBCs for BMT (Investigations) | 6 (6) | 0 (0)
Urinary frequency/urgency (Renal and urinary disorders) | 2 (4) | 0 (0)
Vasovagal episode (Nervous system disorders) | 1 (1) | 0 (0)
Voice changes/stridor/larynx (e.g., hoarseness, loss of voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 8 (11) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0)
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hematologic-Other (Splenomegaly in donor-resolved) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hot flashes/flushes (Vascular disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (4) | 0 (0) — (fever of unknown origin without clinically or microbiologically documented infection)
Diarrhea for BMT (Gastrointestinal disorders) | 3 (4) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No